CLINICAL TRIAL: NCT02944396
Title: A Phase 1 Dose-Escalation and Phase 2 Randomized, Open-Label Study of Nivolumab and Veliparib in Combination With Platinum Doublet Chemotherapy in Subjects With Metastatic or Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Veliparib in Combination With Nivolumab and Platinum Doublet Chemotherapy in Participants With Metastatic or Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-534; 2016-001658-16 (EudraCT Number)
Record Dates: First submitted 2016-10-19; First posted 2016-10-25 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: metastatic; non-small cell lung cancer; Eastern Cooperative Oncology Group (ECOG); veliparib; nivolumab; Platinum Doublet Chemotherapy; carboplatin; paclitaxel; pemetrexed; Response Evaluation Criteria In Solid Tumors (RECIST); Common Terminology Criteria for Adverse Events (CTCAE); Poly (ADP) ribose polymerase (PARP); Immuno Oncology; Metastatic or Advanced Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Pemetrexed; Nivolumab; Paclitaxel; veliparib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Veliparib and nivolumab with platinum doublet chemotherapy (Experimental): Veliparib and nivolumab in combination with platinum doublet chemotherapy (carboplatin/paclitaxel or carboplatin/pemetrexed)
  Interventions: Drug: pemetrexed; Drug: nivolumab; Drug: paclitaxel; Drug: veliparib; Drug: carboplatin
- Veliparib with platinum doublet chemotherapy (Experimental): Veliparib in combination with platinum doublet chemotherapy (carboplatin/paclitaxel or carboplatin/pemetrexed)
  Interventions: Drug: pemetrexed; Drug: paclitaxel; Drug: veliparib; Drug: carboplatin

INTERVENTIONS:
Drug: pemetrexed — intravenous; administered on Day 1 via infusion in a 21-day cycle
  Other Names: Alimta
Drug: nivolumab — intravenous; administered on Day 1 via infusion in a 21-day cycle
  Other Names: Opdivo
  Arms: Veliparib and nivolumab with platinum doublet chemotherapy
Drug: paclitaxel — intravenous; administered on Day 1 via infusion in a 21-day cycle
  Other Names: Taxol
Drug: veliparib — oral capsule; varying doses administered on Days -2 to 5 in a 21-day cycle
  Other Names: ABT-888
Drug: carboplatin — intravenous; administered on Day 1 via infusion in a 21-day cycle
  Other Names: Paraplatin

SUMMARY:
This study seeks to establish the recommended Phase 2 dose (RPTD) of veliparib in combination with nivolumab and platinum doublet chemotherapy (carboplatin/paclitaxel or carboplatin/pemetrexed) (Phase 1 portion) and to assess whether the addition of nivolumab to veliparib in combination with platinum doublet chemotherapy results will improve progression free survival (PFS) compared to veliparib with platinum doublet chemotherapy alone in participants with metastatic or advanced Non-small Cell Lung Cancer (NSCLC) (Phase 2 portion).

A strategy decision was made not to proceed to Phase 2 portion of this study due to change in standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a life expectancy greater than 12 weeks,
* Participant must have cytologically or histologically confirmed Non-small Cell Lung Cancer (NSCLC).
* Participant must have metastatic or advanced NSCLC (Stage IIIB or IV) that is not amenable to surgical resection or radiation or chemoradiation with curative intent at time of study screening.
* Participant must have at least 1 unidimensional measurable NSCLC lesion on a computed tomography (CT) scan as defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1).
* Participant must have resolution to Grade 1 or lower of any toxic effects (excepting alopecia) of the most recent therapy prior to Cycle 1 Day 2.
* Participant must have an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 to 1.
* Participant must have adequate bone marrow, renal, and hepatic function.

Exclusion Criteria:

* Participant has received prior cytotoxic chemotherapy (including chemotherapy in combination with radiotherapy) for NSCLC, except for adjuvant or neoadjuvant therapy accompanied by surgery with curative intent that was completed one year prior to Cycle 1 Day -2.
* Participant has received prior therapy with a Poly-(ADP-ribose)-Polymerase (PARP) inhibitor.
* Participant has received prior treatment with any anti-programmed cell death protein-1 (anti-PD-1), or PD Ligand-1 (PD-L1) or PD Ligand-2 (PD-L2) agent or an antibody targeting other immunoregulatory receptors or mechanisms.
* Participant has received radiation therapy to lung greater than 30 Gy within 6 months, or antineoplastic biologic therapy within 21 days, or major surgery within 21 days, or tyrosine kinase inhibitor therapy within 7 days, or palliative radiation within 7 days of the first dose of study medication.
* Participant has untreated central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 3.5 years
  PFS is defined as the number of days from the date of randomization to the date of earliest disease progression (radiographic progression per RECIST version 1.1 or clinical disease progression) or death. If the participant does not experience disease progression or death, then the data will be censored at the date of the last disease assessment.
Recommended Phase 2 dose (RPTD) of veliparib (ABT-888) in combination with nivolumab and platinum doublet chemotherapy in participants with metastatic or advanced Non-Small Cell Lung Cancer (NSCLC). | Up to 6 weeks

SECONDARY OUTCOMES:
Tmax for pemetrexed | Up to approximately 3 weeks
AUC for nivolumab | Up to approximately 3.5 years
Overall Survival (OS) | Up to approximately 3.5 years
  OS is defined as the number of days from the date of randomization to the date of death. For subjects who did not die, their data will be censored at the date of last study visit or the last known date to be alive, whichever is later.
Tmax for nivolumab | Up to approximately 3.5 years
AUC for pemetrexed | Up to approximately 3 weeks
Time to Cmax (peak time, Tmax) for veliparib | Up to approximately 9 weeks
Area under the plasma concentration-time curve (AUC) for veliparib | Up to approximately 9 weeks
Maximum observed serum concentration (Cmax) of nivolumab anti-drug antibody (ADA) | Up to approximately 3.5 years
Duration of Overall Response (DOR) | Up to approximately 3.5 years
  DOR is defined as the number of days from the date of first response (CR or PR) to the earliest documentation of progressive disease or death due to disease progression.
Maximum observed plasma concentration (Cmax) for pemetrexed | Up to approximately 3 weeks
Maximum observed plasma concentration (Cmax) for veliparib | Up to approximately 9 weeks
Objective Response Rate (ORR) | Up to approximately 3.5 years
  ORR is defined as the proportion of the participants who have a complete response (CR) or partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (6):
- United States (6):
  - University of Alabama at Birmingham - Main /ID# 155135, Birmingham, Alabama
  - Icri /Id# 155593, Whittier, California
  - Univ of Colorado Cancer Center /ID# 153820, Aurora, Colorado
  - University of Chicago /ID# 153824, Chicago, Illinois
  - Goshen Center for Cancer Care /ID# 153822, Goshen, Indiana
  - Duke University Medical Center /ID# 153821, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No